CLINICAL TRIAL: NCT06955377
Title: Effect of Forward Trunk Flexion in Patients With Parkinson's Disease on the Airway Defense System
Brief Title: Effect of Trunk Flexion on Airway Defense in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Kateřina Dvořáková, Physiotherapist, General University Hospital, Prague
Other Study IDs: 16/25 S-IV
Record Dates: First submitted 2025-04-22; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Postural abnormalities; Airway defense system
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Parkinson's disease: Participants of both groups will attend a total of five visits. During each visit, the participants will undergo a complete assessment including respiratory muscle strength, cough strength, dynamic spirometry, grip strength via a digital hand dynamometer, and evaluation of pulmonary dysfunction using the Index of Pulmonary Dysfunction (IPD) questionnaire. Each examination will last approximately 20 minutes, with no specific training or additional procedures required between visits.
- Patients with Parkinson's disease and forward trunk flexion: Patients with pathological forward trunk flexion defined as thoracic (≥25°) or lumbar flexion (>15°) in standing and walking, which completely disappears in the supine position.
  Participants of both groups will attend a total of five visits. During each visit, the participants will undergo a complete assessment including respiratory muscle strength, cough strength, dynamic spirometry, grip strength via a digital hand dynamometer, and evaluation of pulmonary dysfunction using the Index of Pulmonary Dysfunction (IPD) questionnaire. Each examination will last approximately 20 minutes, with no specific training or additional procedures required between visits.

SUMMARY:
The main mechanisms of airway protection include a properly functioning swallowing process and a cough. Studies focusing on patients with Parkinson's disease (PD) have previously demonstrated impairments in both swallowing (dysphagia) and coughing (dystussia). Aspiration pneumonia is the leading cause of death in individuals with PD.

Swallowing function is directly related to body posture. Postural abnormalities (PA) are a common symptom of PD and significantly contribute to patient disability, affect respiratory function, and reduce quality of life. Previous research has shown that more than 20% of PD patients suffer from some form of PA.

Most PD patients with a forward trunk flexion angle greater than 30 degrees report specific difficulties, such as dysphagia. A link has previously been demonstrated between postural abnormalities associated with flexed posture and restrictive ventilatory impairment. It can be assumed that this restrictive ventilatory impairment, which reduces the amount of air the patient can inhale into the lungs and subsequently exhale, negatively affects the strength of voluntary cough. However, this hypothesis has not yet been verified in the mentioned patient group.

The primary aim of the study will be to examine the effect of forward trunk flexion (FTF) in Parkinson's disease on the airway defense system.

DETAILED DESCRIPTION:
The primary aim of the study will be to verify the potential relationship between forward trunk flexion, respiratory muscle strength, and the strength of voluntary cough.

Hypotheses:

1. Forward trunk flexion in patients with Parkinson's disease (PD) will negatively affect respiratory muscle strength and the strength of voluntary cough.
2. Respiratory muscle strength and the strength of voluntary cough will deteriorate more rapidly over a three-year period in patients with PD and forward trunk flexion than in patients with PD without forward trunk flexion.

The secondary aim will be to correlate respiratory muscle strength and the strength of voluntary cough with handgrip strength and the pulmonary dysfunction index as potential screening methods.

Hypothesis:

1. Handgrip strength and the pulmonary dysfunction index will correlate with respiratory muscle strength and the strength of voluntary cough.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson' s disease
* Age ≥ 18 years

Exclusion Criteria:

* Unreliable performance of MIP, MEP, or grip strength measurements, for example, due to cognitive deficits (assessed by the researcher)
* Inadequate lip seal
* Significant deformities of the dominant hand that could affect the accuracy of grip strength measurements
* Other severe neurological diseases apart from PD
* History of unstable cardiovascular disease
* Severe pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study, participants will be selected from patients with Parkinson's Disease who are being monitored at the Extrapyramidal Center of the Neurology Clinic and the Center for Clinical Neuroscience at the First Faculty of Medicine, Charles University, and the General University Hospital in Prague.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Voluntary peak cough flow | baseline, 12months, 24months, 36months
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.
Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) | baseline, 12months, 24months, 36months
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.
Forced vital capacity (FVC) | baseline, 12months, 24months, 36months
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.
Forced expiratory volume (FEV1) | baseline, 12months, 24months, 36months
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.
Peak expiratory flow (PEF) | baseline, 12months, 24months, 36months
  Assessments will be performed in accordance with American Thoracic Society/European Thoracic Society guidelines.

SECONDARY OUTCOMES:
Hand grip strength | baseline, 12months, 24months, 36months
  The assessment of hand grip strength will be conducted according to the recommendations of the American Society of Hand Therapists. A digital hand dynamometer will be used.
Index of Pulmonary Dysfunction (IPD) | baseline, 12months, 24months, 36months
  The screening assessment using the IPD questionnaire will involve the evaluation of four clinical indicators. The first two are direct questions asked to the patient regarding mucus management and cough strength. The third item is the strength of the voluntarily induced cough, subjectively assessed by the examiner. The fourth item tests the patient's ability to count out loud for as long as possible after a maximum inspiratory effort.

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Forsyth AL, Joshi RY, Canning CG, Allen NE, Paul SS. Flexed Posture in Parkinson Disease: Associations With Nonmotor Impairments and Activity Limitations. Phys Ther. 2019 Jul 1;99(7):893-903. doi: 10.1093/ptj/pzz033. PMID 30830153
- [Background] Margraf NG, Granert O, Hampel J, Wrede A, Schulz-Schaeffer WJ, Deuschl G. Clinical Definition of Camptocormia in Parkinson's Disease. Mov Disord Clin Pract. 2016 Oct 11;4(3):349-357. doi: 10.1002/mdc3.12437. eCollection 2017 May-Jun. PMID 30363363
- [Background] Tinazzi M, Gandolfi M, Ceravolo R, Capecci M, Andrenelli E, Ceravolo MG, Bonanni L, Onofrj M, Vitale M, Catalan M, Polverino P, Bertolotti C, Mazzucchi S, Giannoni S, Smania N, Tamburin S, Vacca L, Stocchi F, Radicati FG, Artusi CA, Zibetti M, Lopiano L, Fasano A, Geroin C. Postural Abnormalities in Parkinson's Disease: An Epidemiological and Clinical Multicenter Study. Mov Disord Clin Pract. 2019 Jun 29;6(7):576-585. doi: 10.1002/mdc3.12810. eCollection 2019 Sep. PMID 31538092
- [Background] Claus I, Muhle P, Czechowski J, Ahring S, Labeit B, Suntrup-Krueger S, Wiendl H, Dziewas R, Warnecke T. Expiratory Muscle Strength Training for Therapy of Pharyngeal Dysphagia in Parkinson's Disease. Mov Disord. 2021 Aug;36(8):1815-1824. doi: 10.1002/mds.28552. Epub 2021 Mar 2. PMID 33650729
- [Background] Troche MS, Curtis JA, Sevitz JS, Dakin AE, Perry SE, Borders JC, Grande AA, Mou Y, Vanegas-Arroyave N, Hegland KW. Rehabilitating Cough Dysfunction in Parkinson's Disease: A Randomized Controlled Trial. Mov Disord. 2023 Feb;38(2):201-211. doi: 10.1002/mds.29268. Epub 2022 Nov 7. PMID 36345090